CLINICAL TRIAL: NCT04753099
Title: A Randomized Control Pilot Study to Examine the Effectiveness of Telehealth Occupation-Based Coaching for Families With a Child With Type 1 Diabetes
Brief Title: Telehealth Family Coaching With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Vanessa Jewell, Principal Investigator, Creighton University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Telehealth Coaching
Record Dates: First submitted 2020-09-09; First posted 2021-02-15 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receives occupation-based coaching via telehealth
  Interventions: Behavioral: occupation-based coaching
- Control (No Intervention): No intervention Will receive the occupation-based coaching via telehealth after the 12-weeks

INTERVENTIONS:
Behavioral: occupation-based coaching — Occupation based coaching is an intervention proven to be an effective intervention in family-centered practice. OBC is a strength-based approach that emphases collaboration with clients in goals setting and attainment to increase overall health and quality of life. Clients are the central focus of the intervention and generate their own strategies to address goals as part of the coaching process. In their role as coach, the therapists employ techniques such as reflective questioning and comments to support clients in identifying existing routines and rituals that impact goal attainment and to increase knowledge and access to resources that can promote improved caregiver quality of life after a child's diagnoses with T1D. Occupation based coaching can be divided into the following steps: "(1) setting goals, (2) exploring options, (3) planning action, (4) carrying out the plan, (5) checking performance, and (6) generalizing"(Little et al., 2018, p.2).
  Other Names: family coaching
  Arms: Intervention

SUMMARY:
Telehealth is a delivery format that shows promise, and occupation-based coaching (OBC) is one intervention that can be delivered via telehealth. OBC is a collaborative coaching model with the therapist and the family (caregiver and child) that has been shown to improve positive child-caregiver interactions, caregiver competence with managing child health maintenance tasks, and improve engagement in meaningful everyday tasks (such as health maintenance tasks, self-care, and social participation). The goal of this pilot study is to improve child health outcomes and family quality of life for young children diagnosed with type 1 diabetes. Specifically, this pilot randomized control trial will provide valuable information about the preliminary effectiveness of occupation-based coaching (OBC) via telehealth to improve the quality of life of families and children diagnosed with type 1 diabetes (T1D). It is hypothesized that OBC is an effective intervention that can be delivered to T1D families living in rural communities via telehealth methods.

DETAILED DESCRIPTION:
Design The research investigators plan to use a randomized control trial design with a small sample size (n=16) to gather pilot data. This pilot data will provide the foundation for a future full-scale clinical trial.

This study utilizes Occupation-Based-Coaching (OBC) via telehealth to improve quality of life of families and children diagnosed with type 1 diabetes living in rural communities. Occupation based coaching is an intervention founded on the principles of occupational performance coaching and has proven to be an effective intervention in family-centered practice. OBC is a strength-based approach that emphases collaboration with clients in goals setting and attainment to increase overall health and quality of life. Clients are the central focus of the intervention and generate their own strategies to address goals as part of the coaching process. In their role as coach, the therapists employ techniques such as reflective questioning and comments to support clients in identifying existing routines and rituals that impact goal attainment and to increase knowledge and access to resources that can promote improved caregiver quality of life after a child's diagnoses with T1D. Occupation based coaching can be divided into the following steps: "(1) setting goals, (2) exploring options, (3) planning action, (4) carrying out the plan, (5) checking performance, and (6) generalizing." An expert in occupation-based coaching will provide intervention protocol training to the research team. An intervention fidelity measure, providing more information about the intervention, is attached as an Addendum.

Procedure Participants will be recruited through use of social media platforms, ResearchMatch, snowball sampling /referrals, and Juvenile Diabetes Research Foundation outreach events. Written consent from the guardian, assent from children aged 7-12, and parental permission forms will be obtained prior to the beginning the study. Through simple randomization, 16 families (caregiver/child dyads) will be allocated into either the control group or the intervention group. Due to IRB regulations and ethics, the control group will receive the intervention after study completion. A research team member will then call the guardian to schedule the CGM training, evaluation, and the first intervention appointment (if in the intervention group). Each subsequent visit and post-evaluation will be scheduled the week prior.

Prior to starting the intervention, participants in the control and intervention group will receive training regarding continuous glucose monitor (CGM) from a certified diabetes educator. The CDE will deliver the training in a group setting as able (individual if needed due to scheduling or participant preference) via Zoom, the training will last approximately 60-90 minutes. If the participants were previously using a Dexcom, the training will likely be shorter at 30-60 minutes. The training will be followed by a two-week trial with the CGM to ensure comfort and competence using the CGM device.

After the trial period is concluded, the team evaluators (registered nurse, registered occupational therapist) will administer all assessments. The registered nurse will administer the Demographic Family Form (2-3 minutes) with the caregiver, WHO-QOL (10 minutes) with the caregiver, and provide directions for the at-home hemoglobin a1c testing (5 minutes) with the caregiver and child. Procedures for the hemoglobin a1c are outlined in an addendum. The occupational therapist evaluator will administer the Parental Scale of Competence (5 minutes) with the caregiver and Goal Attainment Scale (5-10 minutes) with the caregiver and child as appropriate. Time-in-Range will be read separately from the CGM application, and the certified diabetes educator will pull all data from the application. The CGM reads the child's blood glucose levels. Approximately 30 minutes total will be allocated for the evaluation. All evaluators are blinded to the group assignments to decrease risk of bias. The study participants will have access to the certified diabetes educator to ask questions about the CGM throughout the study.

After the two-week trial with the CGM, the families will begin the 12-weeks of either receiving the intervention/OBC or control/standard care. During the 12 weeks, the control group will receive standard care (Table 1) for a child with type 1 diabetes continued by their current medical provider.

The intervention group will receive occupation-based-coaching via telehealth, along with standard care. Individual intervention sessions will be conducted 1 time per week for a 1-hour period by a licensed occupational therapy practitioner and /or student supervised by a licensed occupational therapy practitioner. The intervention will be delivered via telehealth, utilizing a private room equipped with telehealth technology. Telehealth intervention will be provided through Zoom for HealthCare, a Health Insurance Portability and Accountability Act of 1996 (HIPAA) compliant video platform. Prior to each session, families will receive an email with a link to connect to the teleconference and a text reminder the day before the scheduled session. After completion of a 12-week intervention period, outcome measures will be re-administered by the nurse and/or occupational therapy practitioner, who remains blinded to participants' group allocation. All sessions will be recorded via Zoom and saved on the research computer. The recorded sessions will be sent to rev.com or other comparable transcription service for transcription. The evaluators will then code the transcriptions for intervention fidelity.

A research team evaluator will administer all outcome measures and will be blinded to the intervention and control group to ensure rigor and avoid bias. All family member participants will be given a unique, anonymous identifier to maintain confidentiality. The research team will store all documents and data in a shared OneDrive (a secure cloud drive) that is only accessible to the research team and will keep the data for 3 years after study completion, per IRB guidelines. The research team completed all CITI training modules and are received additional training on adverse and unexpected events from the IRB office prior to starting the study. The researchers will immediately report any adverse or unexpected events to the IRB office and fill out the appropriate forms.

ELIGIBILITY:
Inclusion Criteria:

* caregivers and children diagnosed with type 1 diabetes
* one hour commute to pediatric endocrinology office
* reside in NE, IA, MN, or CO
* caregiver must be 19 years old or older

Exclusion Criteria:

* child is currently receiving occupational therapy services

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Quality of Life survey to measure physical health, psychological health, social relationships, and environmental health. | A change from baseline to 12 weeks
  This survey is a 26-item instrument consisting of four domains: physical health, psychological health, social relationships, and environmental health. This survey is also contains quality of life and general health items. Each individual item is scored from 1 to 5 on a response scale (1 being low and 5 being high).
family-centered participation goals | A change from baseline to 12 weeks
  Goal Attainment Scale measures whether goals are met or not on a scale of (-2 being much worse than the current situation to +2 being much better than the current situation.
time-in-range | A change from baseline to 12 weeks
  continuous glucose monitor
hemoglobin a1c number | A change from baseline to 12 weeks
  biometric
parental competence with managing child's care | A change from baseline to 12 weeks
  Parenting Sense of Competence Scale. Parent's rate 17 items on a scale of 1-6 (1 meaning strongly disagree and 6 meaning strongly agree). A higher total score indicates a higher parenting sense of competency. There are no average scores or 'cut-off's' for this tool.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Jewell, PhD, OTR/L, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cason J, Behl D, Ringwalt S. Overview of States' Use of Telehealth for the Delivery of Early Intervention (IDEA Part C) Services. Int J Telerehabil. 2012 Dec 9;4(2):39-46. doi: 10.5195/IJT.2012.6105. eCollection 2012 Fall. PMID 25945202
- [Background] Little LM, Pope E, Wallisch A, Dunn W. Occupation-Based Coaching by Means of Telehealth for Families of Young Children With Autism Spectrum Disorder. Am J Occup Ther. 2018 Mar/Apr;72(2):7202205020p1-7202205020p7. doi: 10.5014/ajot.2018.024786. PMID 29426380
- [Background] Zylstra, S.E. (2013). Evidence for the use of telehealth in pediatric occupational therapy. Journal of Occupational Therapy, Schools, and Early Intervention, 6, 326-355.
- [Background] Graham F, Rodger S, Ziviani J. Coaching parents to enable children's participation: an approach for working with parents and their children. Aust Occup Ther J. 2009 Feb;56(1):16-23. doi: 10.1111/j.1440-1630.2008.00736.x. PMID 20854485